CLINICAL TRIAL: NCT02649062
Title: Study of the Pharmacodynamics of NGM282 on Colonic Transit, Bile Acid Homeostasis, and Fecal Fat in Subjects With Functional Constipation and Healthy Individuals
Brief Title: Study of NGM282 in Subjects With Functional Constipation and Healthy Individuals
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0107
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Functional Constipation
MeSH Terms: interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NGM282 Dose 1 (Experimental): NGM282
  Interventions: Biological: NGM282
- NGM282 Dose 2 (Experimental): NGM282
  Interventions: Biological: NGM282
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NGM282
  Arms: NGM282 Dose 1; NGM282 Dose 2
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of NGM282 on colonic transit, bile acid homeostasis, and fecal fat in subjects with functional constipation and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Functional constipation confirmed by modified Rome III criteria or Healthy Volunteer

Exclusion Criteria:

* Structural or metabolic diseases/conditions that affect the GI system
* Diagnosis of dyspepsia, IBS, or significant gastrointestinal symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Effect on Colon Transit, as measured by the movement of food through the colon | 9 days

SECONDARY OUTCOMES:
Clinical Laboratory Assessments | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Rossi, PharmD, Study Director — NGM Biopharmaceuticals, Inc
Locations (1):
- NGM Clinical Study Site 1, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No